CLINICAL TRIAL: NCT02827383
Title: Pilot Study to Test the Effect of Fractionalized Vigorous-Intensity Activity on Acute Glucose in Adults at Risk for Type 2 Diabetes
Brief Title: Pilot Stair Climbing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Gay (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor-Investigator, Jennifer Gay, Assistant Professor, University of Georgia
Organization: University of Georgia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ID#STUDY00002685
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stair Climbing 4x/day (Experimental): Participants use the stair climber 4 times per day, for 4 minutes at a time. Total dose = 16 minutes.
  Interventions: Behavioral: Stair Climbing Frequency
- Stair Climbing 8x/day (Experimental): Participants use the stair climber 8 times per day, for 2 minutes at a time. Total dose = 16 minutes.
  Interventions: Behavioral: Stair Climbing Frequency

INTERVENTIONS:
Behavioral: Stair Climbing Frequency — Includes 1 sedentary day prior to completing crossover phases.

SUMMARY:
This pilot study seeks to demonstrate feasibility to conduct data collection and illustrate potential for effect of fractionalized bouts of stair climbing on glucose control in adults at risk for type 2 diabetes.

DETAILED DESCRIPTION:
Objective: Compare the short-term effects of two different fractionalized stair climbing bout protocols on glucose control among adults at risk for type 2 diabetes.

Rationale: Fractionalized physical activity is associated with reduced BMI, glycated hemoglobin, lower 2-hr plasma glucose and insulin sensitivity in cross-sectional studies. Yet, few studies have examined the effects of fractionalized or intermittent physical activity in a prospective manner. Furthermore, the research is limited to patients with diagnosed type 2 diabetes, or using exercise of a moderate intensity.

The hypothesis is that stair climbing, a vigorous-intensity activity, may have a greater health effect. However, this has not been tested in short bouts of activity that are spread out during a day.

Implications: Fractionalized physical activity may be more feasible for adults at risk for, or with diagnosed type 2 diabetes who are not currently active. These short bouts can increase energy expenditure throughout the day, rather than in one long continuous bout as currently recommended.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 40 years but less than 65 years (working age adult with reduce physiologic capacity to regulate glucose)
* BMI of overweight or obese (25.0 to 35.0)
* Answered "No" to all questions on the Physical Activity Readiness Questionnaire, or has physician approval to participate
* Hemoglobin A1C% value in the at-risk range of 5.7 to 6.4

Exclusion Criteria:

* Unable to physically perform stair climbing
* Currently exercising for 60 or more minutes weekly.
* Weight over 275 lbs (because stair climbing machine has a weight limit)

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Continuous Glucose Monitor | Up to 5 days
  Participant has device inserted prior to dinner the night before the sedentary day, completes the sedentary day and two stair climbing days, then has the device removed on the morning of the 5th day.

SECONDARY OUTCOMES:
Heart Rate | 2 Intervention Days
  Measuring heart rate during stair climbing for % max heart rate and % heart rate reserve. Heart rate will be measured during the stair climbing bouts on each of the two intervention days.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Gay, PhD, Principal Investigator — University of Georgia
Locations (1):
- Clinical and Translational Research Unit, University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is the investigator's intent to make data available after publication of the primary research questions. The method by which data will be made available is yet to be determined.

REFERENCES:
- [Derived] Gay JL, Buchner DM, Erickson ML, Lauture A. Effect of short bouts of high intensity activity on glucose among adults with prediabetes: A pilot randomized crossover study. Diabetes Res Clin Pract. 2018 Jul;141:168-174. doi: 10.1016/j.diabres.2018.04.045. Epub 2018 May 7. PMID 29746878